CLINICAL TRIAL: NCT01347866
Title: A Multi-arm Phase 1 Dose Escalation Study Of The Safety, Pharmacokinetics, And Pharmacodynamics Of The Dual Pi3k/Mtor Inhibitors Pf-04691502 And Pf-05212384 In Combination With Experimental Or Approved Anticancer Agents In Patients With Advanced Cancer
Brief Title: Clinical Study Of PI3K/mTOR Inhibitors In Combination With An Oral MEK Inhibitor Or Irinotecan In Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Refer to Detailed Description for documentaion of Termination Statement.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Basic Science
Other Study IDs: B1271002; 2011-001671-39 (EudraCT Number)
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-02

CONDITIONS: Advanced Cancer
Keywords: Advanced metastatic cancer (solid tumors); PI3K; mTOR; MEK
MeSH Terms: interventions — gedatolisib; mirdametinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm D: PF-05212384 + PD-0325901 (Experimental)
  Interventions: Drug: PF-05212384; Drug: PD-0325901
- Arm C: PF-05212384 + irinotecan (Experimental)
  Interventions: Drug: PF-05212384; Drug: irinotecan

INTERVENTIONS:
Drug: PF-05212384 — PF-05212384 intravenous infusion weekly starting at 110 mg.
  Arms: Arm D: PF-05212384 + PD-0325901
Drug: PD-0325901 — PD-0325901 Oral twice daily (BID) dosing 2 mg BID 3 weeks on 1 week off
  Arms: Arm D: PF-05212384 + PD-0325901
Drug: PF-05212384 — PF-05212384 intravenous infusion weekly starting at 95 mg.
  Arms: Arm C: PF-05212384 + irinotecan
Drug: irinotecan — Irinotecan by intravenous infusion at 180 mg/m2 every two weeks (Q x 2 week)
  Arms: Arm C: PF-05212384 + irinotecan

SUMMARY:
After the fourth protocol amendment two study arms are evaluated in this clinical protocol: PD-0325901 (oral MEK inhibitor) plus PF-05212384 (intravenous PI3K/mTOR inhibitor) and PF-05212384 plus irinotecan. The study will assess safety, pharmacokinetics and pharmacodynamics of these combinations in patients with advanced cancer. Once the maximum tolerated doses are identified, further assessment of these combinations will be done in patients with previously treated metastatic colorectal or pancreatic cancer for the PF-05212384 plus irinotecan arm and in patients with ovarian cancer or KRAS mutated non small cell lung cancer for the combination of PF-05212384 plus PD-0325901.

DETAILED DESCRIPTION:
The study was prematurely discontinued as a result of an internal portfolio review on April 1, 2015. The decision to terminate was not due to any safety or efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced/metastatic solid tumor for which there is no currently clinically effective treatment.
* All tumor types for patients enrolled in Stage 1 of Arm C.
* For patients enrolled in Stage 2 of Arm C, advanced colorectal cancer (both KRAS mutated and KRAS wild type), which has progressed on irinotecan-based regimens, and pancreatic ductal adenocarcinoma after progression on first line treatment for metastatic/advanced disease.
* For patients enrolled in Stage 1 of Arm D, tumors with KRAS or BRAF mutation (archived or fresh biopsy). Patients with tumors harboring other mutations that activate the MAPK pathway may be enrolled upon agreement with the Sponsor.
* For patients enrolled in Stage 2 of Arm D, ovarian cancer which has progressed on prior platinum containing regimen or KRAS mutated non small cell lung cancer which has progressed on one prior regimen.
* Patients with colorectal cancer enrolled to both Arms must:

  1. have received at least 6 weeks of irinotecan-based therapy (either as single agent or in combination with cytotoxic drugs or in combination with targeted therapies) as the last prior treatment
  2. have progressed on or within 1 month of completing this irinotecan-based regimen
* All patients must provide an archived or fresh tumor sample.
* For a subset of patients fresh tumor biopsies are mandatory:

  a. All patients with CRC enrolled to Stage 2 of Arm C must provide a fresh tumor biopsy at baseline. A subset of patients (10 or more) with at least 5 evaluable patients with CRC KRAS wild type must also provide tumor biopsy during treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) must be 0 or 1
* Adequate Bone Marrow, Renal, Cardiac, and Liver Function

Exclusion Criteria:

* -Patients with known active brain metastases
* -Chemotherapy, radiotherapy (other than palliative radiotherapy to lesions that will not be followed for tumor assessment on this study, ie, non target lesions), biological or investigational agents within 4 weeks of the start of the study treatment (6 weeks for mitomycin C or nitrosoureas).
* -Any surgery (not including minor procedures such as lymph node biopsy, needle biopsy, and/or placement of port-a-cath) within 4 weeks of start of the study treatment; or not fully recovered from any side effects of previous procedures.
* -In Arm D only: Patients with glaucoma, intraocular pressure > 21 mmHg, history of retinal vein occlusions, ocular ischemia or any other clinically significant abnormality in the ophthalmologic exam which would make the patient inappropriate for entry into this study
* -For patients enrolling in Stage 2 prior therapy with an agent that is known or proposed to be active by action on PI3K and/or mTOR.
* -Prior high dose chemotherapy requiring hematopoietic stem cell transplantation within 12 months of study treatment start.
* -Known impaired pulmonary function or demonstrated to be impaired by Pulmonary Function Test (PFT) for patients who present with clinical suggestion of impairment.
* -Uncontrolled or significant cardiovascular disease
* -Current use or anticipated need for food or drugs that are known potent CYP3A4 inhibitors
* - Current or anticipated need for food or drugs that are known potent CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (14):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UCLA Oncology Center, Los Angeles, California
  - Santa Monica - UCLA Medical Center and Orthopaedic Hospital, Santa Monica, California
  - UCLA Santa Monica Hematology Oncology, Santa Monica, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Denver (CTRC), Aurora, Colorado
  - University of Colorado Hospital Anschutz Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC, Investigational Drug Services, Charleston, South Carolina
  - MUSC Health East Cooper, Mt. Pleasant, South Carolina
  - MUSC Specialty Care-North, North Charleston, South Carolina
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Ospedale San Raffaele, Milan, Italy
- Hospital General Vall d'Hebron, Barcelona, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1271002&StudyName=Clinical%20Study%20Of%20PI3K/mTOR%20Inhibitors%20In%20Combination%20With%20An%20Oral%20%20MEK%20Inhibitor%20Or%20Irinotecan%20In%20Patients%20With%20Advanced%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Arms A and B, 7 and 14 participants were screed and received study treatment, respectively. In Arm C, 45 participants were screened and 44 received study treatment. In Arm D, 39 participants were screened and 37 received study treatment. There was no Stage 2 for Arm D, the study was terminated before enrolling patients to Stage 2 for Arm D.
Groups:
- PF-04691502+PF-0325901: Arm A1 (Stage1): Single oral dose of PF-04691502 4 mg tablet and PF 0325901 8 mg capsule in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 4 mg tablet orally once daily and PF 0325901 8 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-04691502+PF 0325901: Arm A2 (Stage1): Single oral dose of PF-04691502 6 mg tablet and PF 0325901 8 mg capsule in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 6 mg tablet orally once daily and PF 0325901 8 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-04691502+PF 0325901: Arm A4 (Stage1): Single oral dose of PF-04691502 4 mg tablet and PF 0325901 5 mg capsule in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 4 mg tablet orally once daily and PF 0325901 5 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-04691502+Irinotecan: Arm B1 (Stage 1): Single oral dose of PF-04691502 4 mg tablet in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 4 mg tablet orally once daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death. Irinotecan 180 mg/m^2 dosed intravenously biweekly.
- PF-04691502+Irinotecan: Arm B2 (Stage 1): Single oral dose of PF-04691502 6 mg tablet in lead-in period (4 to 10 days prior to Cycle 1 Day 1), followed by PF-04691502 6 mg tablet orally once daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death. Irinotecan 180 mg/m^2 dosed intravenously biweekly.
- PF-05212384+Irinotecan: Arm C1 (Stage 1): Participants received intravenous doses of PF-05212384 95 mg weekly on Days 2, 9, 16 and 23 of each 28 day cycle. Irinotecan 180 mg/m^2 dosed intravenously biweekly.
- PF-05212384+Irinotecan: Arm C2 (Stage 1): Participants received intravenous doses of PF-05212384 110 mg weekly on Days 2, 9, 16 and 23 of each 28 day cycle. Irinotecan 180 mg/m^2 dosed intravenously biweekly.
- PF-05212384+Irinotecan: Arm C3 (Stage 1): Participants received intravenous doses of PF-05212384 130 mg weekly on Days 2, 9, 16 and 23 of each 28 day cycle. Irinotecan 180 mg/m^2 dosed intravenously biweekly.
- PF-05212384+Irinotecan: Arm C2 (Stage 2): Participants received intravenous doses of PF-05212384 110 mg weekly on Days 2, 9, 16 and 23 of each 28 day cycle. Irinotecan 180 mg/m^2 dosed intravenously biweekly. During Stage 2, only participants with metastatic colorectal cancer (mCRC) and pancreatic ductal adenocarcinoma (PDAC) were enrolled.
- PF-05212384+ PD-0325901: Arm D0 (Stage 1): Single intravenous dose of PF-05212384 110 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 110 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 2 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF-0325901 2 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+ PD-0325901: Arm D0A (Stage 1): Single intravenous dose of PF-05212384 130 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 130 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 2 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF-0325901 2 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+ PD-0325901: Arm D0B (Stage 1): Single intravenous dose of PF-05212384 154 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 154 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 2 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF 0325901 2 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+PD-0325901: Arm D1 (Stage 1): Single intravenous dose of PF-05212384 110 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 110 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 4 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF-0325901 4 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+ PD-0325901: Arm D1A (Stage 1): Single intravenous dose of PF-05212384 130 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 130 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 4 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF-0325901 4 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+PD-0325901: Arm D1B (Stage 1): Single intravenous dose of PF-05212384 154 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 154 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 4 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF-0325901 4 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+ PD-0325901: Arm D2 (Stage 1): Single intravenous dose of PF-05212384 110 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 110 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 6 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF-0325901 6 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+ PD-0325901: Arm D2A (Stage 1): Single intravenous dose of PF-05212384 130 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 130 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 6 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF-0325901 6 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
Period: Overall Study
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+ PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Started | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 4 | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 3 | 1 | 1 | 4 | 5 | 0 | 5 | 3 | 22 | 5 | 0 | 3 | 4 | 4 | 2 | 3 | 0
Not completed — Subject refused further follow-up | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- PF-05212384+ PD-0325901: Arm D1 (Stage 1): Single intravenous dose of PF-05212384 110 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 110 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 4 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF 0325901 4 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- PF-05212384+ PD-0325901: Arm D1B (Stage 1)): Single intravenous dose of PF-05212384 154 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 154 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 4 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF 0325901 4 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
- Total: Total of all reporting groups
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+ PD-0325901: Arm D1B (Stage 1)) | PF-05212384+ PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1) | Total
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (8.7) | 54.0 (0.0) | 49.0 (0.0) | 53.6 (14.1) | 59.1 (12.9) | 67.0 (3.6) | 60.8 (7.2) | 63.3 (14.5) | 56.7 (12.4) | 63.3 (5.9) | 43.3 (9.1) | 64.0 (8.9) | 55.7 (10.0) | 57.9 (12.9) | 61.3 (14.2) | 60.0 (11.8) | 54.5 (9.2) | 58.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 0 | 5 | 2 | 2 | 2 | 2 | 13 | 3 | 1 | 2 | 3 | 2 | 0 | 2 | 2 | 44
  Male | 2 | 1 | 1 | 2 | 5 | 1 | 4 | 2 | 18 | 4 | 2 | 2 | 4 | 5 | 3 | 2 | 0 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose-Limiting Toxicities (DLTs) in First Cycle (28 Days)
Description: DLT was defined as any of the following hematologic or non-hematologic events which were attributable to the combination study drug and occurring in the first 28-day cycle: 1) Grade 4 neutropenia lasting greater than (>)7 days; 2) Febrile neutropenia (defined as neutropenia greater than or equal to [≥]Grade 3 and a body temperature ≥38.5°C); 3) Grade ≥3 neutropenic infection; 4) Grade 3 thrombocytopenia with bleeding; 5) Grade 4 thrombocytopenia; 6) Grade ≥3 toxicities; 7) Persistent, intolerable toxicities which resulted in failure to deliver at least 75% of doses during the first cycle; 8) Persistent, intolerable toxicities which resulted in delay of start of Cycle 2 by more than 2 weeks of scheduled day; 9) Persistent Grade 3 QTc prolongation (QTc >500 msec) after correction of any reversible causes.
Time Frame: Baseline up to 28 days
Population: All enrolled participants who started treatment and who did not have a major pre-specified treatment deviation in the first cycle of treatment in Stage 1.
Measure: Number; unit: percentage of participants
Groups:
- PF-05212384+PD-0325901: Arm D2 (Stage 1): Single intravenous dose of PF-05212384 110 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 110 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 6 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF 0325901 6 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 5 | 3 | 6 | 4 | 7 | 3 | 4 | 7 | 7 | 3 | 3 | 1
percentage of participants | 40.0 | 0 | 100 | 14.3 | 40.0 | 0 | 0 | 50.0 | 14.3 | 0 | 0 | 14.3 | 14.3 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to End of Treatment (EOT) (within 28 days after last treatment administration)
Population: All enrolled participants who started treatment.
Measure: Number; unit: participants
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
participants
  AEs | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
  SAEs | 2 | 1 | 1 | 2 | 5 | 0 | 0 | 2 | 5 | 3 | 1 | 2 | 4 | 1 | 0 | 1 | 0

3. Secondary Outcome: Number of Participants With Treatment-Emergent AEs (TEAEs) by National Cancer Institute (NCI) Common Terminology Criteria (CTC) for AEs (CTCAE) (Version 4.0) Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs are events which occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs were graded by the NCI CTCAE (Version 4.0).
Time Frame: Baseline up to End of Treatment (EOT) (within 28 days after last treatment administration)
Population: All enrolled participants who started treatment.
Measure: Number; unit: participants
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
participants
  Any AEs, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Any AEs, Grade 2 | 2 | 0 | 0 | 5 | 2 | 3 | 4 | 1 | 10 | 2 | 2 | 2 | 3 | 2 | 1 | 3 | 0
  Any AEs, Grade 3 | 2 | 1 | 1 | 2 | 5 | 0 | 0 | 2 | 10 | 3 | 1 | 1 | 2 | 4 | 2 | 0 | 1
  Any AEs, Grade 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Any AEs, Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Any AEs, Missing or Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AEs, Total | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2

4. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Hematology)
Description: Number of participants with NCI CTCAE (version 4.0) grade 1 to 4 hematological test abnormalities. Hematological tests included platelet count, hemoglobin, and white blood cell (WBC) count with 5- part differential.
Time Frame: Baseline, Days 1, 15, and 23 of Cycle 1, Days 1 and 15 of Cycle 2, Day 1 of Cycle 3 and subsequent cycles, up to End of Treatment (within 28 days of last treatment administration)
Population: All enrolled participants who started treatment.
Measure: Number; unit: participant
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
participant
  Anemia | 5 | 1 | 1 | 5 | 6 | 3 | 6 | 4 | 31 | 6 | 3 | 3 | 7 | 5 | 3 | 3 | 2
  Hemoglobin Increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Lymphopenia | 5 | 1 | 1 | 7 | 7 | 3 | 5 | 3 | 22 | 5 | 1 | 1 | 6 | 6 | 3 | 1 | 1
  Absolute Neutrophils | 1 | 0 | 0 | 3 | 3 | 0 | 2 | 3 | 18 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Platelets | 3 | 0 | 0 | 4 | 2 | 1 | 1 | 3 | 10 | 0 | 0 | 2 | 1 | 3 | 1 | 1 | 1
  White Blood Cells | 3 | 0 | 0 | 5 | 3 | 3 | 3 | 4 | 22 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Coagulation)
Description: Number of participants with NCI CTCAE (version 4.0) grade 1 to 4 coagulation test abnormalities. Coagulation tests included partial thromboplastin time (PTT) and prothrombin time (PT) international normalized ratio (INR).
Time Frame: Baseline, Days 1 and 15 of Cycle 1, Days 1 and 15 of Cycle 2, Day 1 of Cycle 3 and subsequent cycles, up to End of Treatment (within 28 days of last treatment administration)
Population: All enrolled participants who started treatment. N=number of evaluable participants for each parameter.
Measure: Number; unit: participant
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
participant
  PTT (N=5,1,1,7,7,3,6,4,31,7,3,4,7,7,3,4,2) | 2 | 0 | 0 | 2 | 5 | 2 | 0 | 2 | 21 | 2 | 3 | 2 | 2 | 5 | 0 | 3 | 2
  PT INR (N=5,1,1,7,7,3,6,4,30,7,3,4,7,7,3,4,2) | 1 | 0 | 1 | 2 | 5 | 0 | 1 | 2 | 13 | 0 | 1 | 1 | 3 | 2 | 1 | 2 | 0

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Chemistry)
Description: Number of participants with NCI CTCAE (version 4.0) grade 1 to 4 chemistry test abnormalities. Chemistry tests included aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]), serum creatinine, total bilirubin, direct/indirect bilirubin, alkaline phosphatase, chloride, uric acid, phosphorus, calcium, magnesium, potassium, sodium, blood urea nitrogen (BUN) or urea, total protein, albumin, glucose, and insulin.
Time Frame: as for outcome 4
Population: All enrolled participants who started treatment.
Measure: Number; unit: participant
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
participant
  ALT | 3 | 0 | 1 | 2 | 3 | 0 | 3 | 3 | 13 | 3 | 1 | 2 | 5 | 4 | 3 | 1 | 2
  Alkaline phosphatase | 3 | 1 | 1 | 5 | 6 | 1 | 3 | 2 | 22 | 4 | 3 | 4 | 6 | 6 | 3 | 4 | 2
  AST | 4 | 0 | 1 | 3 | 5 | 0 | 3 | 2 | 16 | 4 | 2 | 3 | 5 | 6 | 3 | 3 | 2
  Total bilirubin | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 1 | 3 | 2 | 0 | 2 | 1 | 4 | 1 | 1 | 0
  creatinine | 5 | 1 | 0 | 5 | 6 | 3 | 5 | 3 | 21 | 5 | 2 | 3 | 5 | 2 | 3 | 4 | 2
  hypercalcemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  hyperglycemia | 5 | 1 | 1 | 6 | 6 | 3 | 5 | 3 | 25 | 5 | 2 | 3 | 7 | 7 | 2 | 4 | 2
  hyperkalemia | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
  hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1
  hypernatremia | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  hypoalbuminemia | 3 | 1 | 1 | 3 | 6 | 0 | 3 | 3 | 18 | 3 | 2 | 4 | 6 | 6 | 3 | 2 | 2
  hypocalcemia | 3 | 0 | 1 | 4 | 4 | 1 | 0 | 4 | 13 | 2 | 2 | 3 | 1 | 4 | 1 | 1 | 2
  hypoglycemia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0
  hypokalemia | 2 | 1 | 1 | 2 | 3 | 0 | 0 | 3 | 14 | 3 | 1 | 2 | 3 | 4 | 0 | 2 | 1
  hypomagnesemia | 2 | 0 | 0 | 3 | 4 | 2 | 2 | 1 | 10 | 2 | 1 | 2 | 0 | 2 | 1 | 2 | 1
  hyponatremia | 1 | 1 | 0 | 4 | 3 | 0 | 1 | 3 | 14 | 2 | 2 | 2 | 4 | 3 | 1 | 1 | 1
  hypophosphatemia | 4 | 1 | 0 | 2 | 5 | 0 | 2 | 1 | 8 | 1 | 1 | 1 | 3 | 3 | 0 | 1 | 0

7. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Urinalysis)
Description: Number of participants with NCI CTCAE (version 4.0) grade 1 to 4 urinalysis test abnormalities for urine protein.
Time Frame: as for outcome 5
Population: All enrolled participants who started treatment. Number of participants analyzed=number of evaluable participants for each laboratory parameter.
Measure: Number; unit: participant
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 6 | 7 | 3 | 4 | 2
participant | 2 | 1 | 1 | 6 | 4 | 1 | 3 | 1 | 15 | 3 | 0 | 2 | 5 | 4 | 1 | 2 | 0

8. Secondary Outcome: Number of Participants With Vital Signs Values Meeting Prespecified Criteria
Description: Number of participants with vital signs values meeting prespecified criteria. Criteria defined as: 1) absolute systolic blood pressue (SBP) less than or equal to (<=) 100 millimeter of mercury (mmHg); 2) absolute SBP greater than or equal to (>=) 160 mmHg, 3) SBP maximum increase of >=20 mmHg from baseline; 4) SBP maximum increase of >=40 mmHg from baseline; 5) SBP maximum increase of >=60 mmHg from baseline; 6) absolute diastolic blood pressure (DBP) <=60 mmHg; 7) absolute DBP >=100 mmHg; 8) DBP maximum increase of >=10 mmHg from baseline; 9) DBP maximum increase of >=20 mmHg from baseline; 10) DBP maximum increase of >=30 mmHg from baseline; 11) absolute heart rate (HR) <50 beats per minute (bpm); 12) absolute HR >120 bpm.
Time Frame: as for outcome 4
Population: All enrolled participants who started treatment. N=number of participants evaluated against criteria.
Measure: Number; unit: participants
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
participants
  Criterion 1 (N=5,1,1,7,7,3,6,4,31,7,3,4,7,7,3,4,2) | 1 | 0 | 0 | 4 | 3 | 0 | 1 | 1 | 9 | 2 | 2 | 3 | 1 | 2 | 0 | 1 | 2
  Criterion 2 (N=5,1,1,7,7,3,6,4,31,7,3,4,7,7,3,4,2) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0
  Criterion 3 (N=5,1,1,6,7,3,6,4,31,7,3,3,7,4,3,4,1) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 3 | 1 | 1 | 3 | 0 | 0 | 2 | 0
  Criterion 4 (N=5,1,1,6,7,3,6,4,31,7,3,3,7,4,3,4,1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Criterion 5 (N=5,1,1,6,7,3,6,4,31,7,3,3,7,4,3,4,1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Criterion 6 (N=5,1,1,7,7,3,6,4,31,7,3,4,7,7,3,4,2) | 0 | 0 | 0 | 3 | 3 | 1 | 2 | 1 | 14 | 1 | 2 | 1 | 2 | 3 | 1 | 1 | 1
  Criterion 7 (N=5,1,1,7,7,3,6,4,31,7,3,4,7,7,3,4,2) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion 8 (N=5,1,1,6,7,3,6,4,31,7,3,3,7,4,3,4,1) | 3 | 0 | 1 | 4 | 1 | 1 | 0 | 3 | 10 | 1 | 1 | 2 | 3 | 0 | 1 | 3 | 1
  Criterion 9 (N=5,1,1,6,7,3,6,4,31,7,3,3,7,4,3,4,1) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Criterion10 (N=5,1,1,6,7,3,6,4,31,7,3,3,7,4,3,4,1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Criterion11 (N=5,1,1,7,7,3,6,4,31,7,3,4,7,7,3,4,2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Criterion12 (N=5,1,1,7,7,3,6,4,31,7,3,4,7,7,3,4,2) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0

9. Secondary Outcome: Maximum Plasma Concentrations (Cmax) for PF-05212384 on Cycle 1 Day 2 and Day 16 for Arm C
Time Frame: Cycle 1 Day 2 and Cycle 1 Day 16: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: Enrolled participants treated who had at least 1 of the pharmacokinetic (PK) parameters of interest estimated. N=number of participants contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/milliliter (mL)
Arm/Group | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2)
Number analyzed (Participants) | 2 | 6 | 4 | 30
nanogram (ng)/milliliter (mL)
  Cycle 1 Day 2 (N=2, 6, 4, 30) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 1640 and 3050 ng/mL, respectively. | 3404 (82) | 4759 (25) | 5221 (61)
  Cycle 1 Day 16 (N=3, 6, 4, 28) | 2201 (16) | 2814 (50) | 4656 (32) | 5728 (56)

10. Secondary Outcome: Maximum Plasma Concentrations (Cmax) for PF-05212384 on Cycle 0 Day -14 and Cycle 1 Day 15 for Arm D
Time Frame: Cycle 0 Day -14 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: Enrolled participants treated who had at least 1 of the PK parameters of interest estimated. N=number of participants contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 7 | 3 | 4 | 7 | 6 | 3 | 4 | 2
ng/mL
  Cycle 0 Day -14 (N=7, 3, 4, 7, 6, 3, 4, 2) | 3625 (62) | 5937 (32) | 11170 (16) | 8476 (32) | 8586 (36) | 6279 (70) | 7239 (39) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 9250 and 15200 ng/mL, respectively.
  Cycle 1 Day 15 (N=5, 3, 4, 6, 5, 1, 4, 1) | 8621 (18) | 6153 (34) | 12440 (32) | 8717 (50) | 8913 (54) | 9280 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. | 7989 (45) | 15400 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP.

11. Secondary Outcome: Maximum Plasma Concentrations (Cmax) for PD-0325901 on Cycle 0 Day -1 and Cycle 1 Day 1 for Arm D
Time Frame: Cycle 0 Day -1 and Cycle 1 Day 1: Pre-dose and 1, 2, 4, 6 and 8 hours post-dose.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 7 | 3 | 3 | 7 | 7 | 3 | 3 | 2
ng/mL
  Cycle 0 Day -1 (N=7, 3, 3, 7, 7, 3, 3, 2) | 85.28 (27) | 63.80 (14) | 87.99 (51) | 180.6 (28) | 191.9 (44) | 115.8 (70) | 231.3 (69) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 204 and 372 ng/mL, respectively.
  Cycle 1 Day 1 (N=5, 3, 3, 6, 6, 3, 4, 2) | 91.69 (31) | 74.23 (43) | 64.99 (56) | 138.7 (23) | 183.6 (29) | 114.6 (50) | 211.9 (44) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 247 and 428 ng/mL, respectively.

12. Secondary Outcome: Maximum Plasma Concentrations (Cmax) for PD-0325901 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm A
Time Frame: Cycle 0 Day -7: Pre-dose and 1, 2, 4, 6, 8, 24, and 72 hours post-dose. Cycle 1 Day 12: Pre-dose and 1, 2, 4, 6 and 8 hours post-dose.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
ng/mL
  Cycle 0 Day -7 (N=5, 1, 1) | 304.9 (49) | 280 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 101 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.
  Cycle 1 Day 12 (N=4, 1, 1) | 341.9 (21) | 690 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 182 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

13. Secondary Outcome: Maximum Plasma Concentrations (Cmax) for PF-04691502 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm A
Time Frame: Cycle 0 Day -7 at 0 hours (pre-dose), 1, 2, 4, 6, 8, 24, and 72 hours, and at Cycle 1 Day 12 at 0 hours (pre-dose), 1, 2, 4, 6, 8, and 24 hours.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
ng/mL
  Cycle 0 Day -7 (N=5, 1, 1) | 38.02 (28) | 59.8 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 48.7 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.
  Cycle 1 Day 12 (N=4, 1, 1) | 52.02 (13) | 21.2 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 64.7 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

14. Secondary Outcome: Maximum Plasma Concentrations (Cmax) for PF-04691502 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm B
Time Frame: Cycle 0 Day -7 at 0 hours (pre-dose) and 1, 2, 4, 6, 8, 24, and 72 hours post-dose. Cycle 1 Day 12 at 0 hours (pre-dose), 1, 2, 4, 6 8 and 24 hours post-dose.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1)
Number analyzed (Participants) | 7 | 7
ng/mL
  Cycle 0 Day -7 (N=7, 7) | 41.44 (8.1201) [1 to 8] | 68.41 (31.818) [1 to 4.13]
  Cycle 1 Day 12 (N=7, 5) | 46.81 (19.381) [1 to 4] | 87.30 (37.647) [1.02 to 6]

15. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for PF-05212384 on Cycle 1 Day 2 and Day 16 for Arm C
Time Frame: Cycle 1 Day 2 and Cycle 1 Day 16: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2)
Number analyzed (Participants) | 2 | 6 | 4 | 30
hour (hr)
  Cycle 1 Day 2 (N=2, 6, 4, 30) | 1.30 [1.00 to 1.60] | 1.02 [0.500 to 1.67] | 0.992 [0.500 to 1.00] | 0.500 [0.467 to 1.07]
  Cycle 1 Day 16 (N=3, 6, 4, 28) | 1.00 [1.00 to 1.08] | 0.992 [0.583 to 1.05] | 0.734 [0.500 to 1.00] | 0.525 [0.333 to 2.92]

16. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for PF-05212384 on Cycle 0 Day -14 and Cycle 1 Day 15 for Arm D
Time Frame: Day -14 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 7 | 3 | 4 | 7 | 6 | 3 | 4 | 2
hr
  Cycle 0 Day -14 (N=7, 3, 4, 7, 6, 3, 4, 2) | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 0.983] | 0.500 [0.500 to 0.500] | 0.500 [0.500 to 3.22] | 0.509 [0.500 to 0.583] | 1.00 [0.500 to 3.08] | 0.500 [0.500 to 0.600] | 0.500 [0.500 to 0.500]
  Cycle 1 Day 15 (N=5, 3, 4, 6, 5, 1, 4, 1) | 0.500 [0.500 to 0.500] | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 0.517] | 0.509 [0.500 to 0.567] | 0.517 [0.500 to 0.583] | 0.667 [0.667 to 0.667] | 0.500 [0.500 to 3.92] | 0.500 [0.500 to 0.500]

17. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for PD-0325901 on Cycle 0 Day -1 and Cycle 1 Day 1 for Arm D
Time Frame: Cycle 0 Day -1 and Cycle 1 Day 1: Pre-dose and 1, 2, 4, 6 and 8 hours post-dose.
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 7 | 3 | 3 | 7 | 7 | 3 | 3 | 2
hr
  Cycle 0 Day -1 (N=7, 3, 3, 7, 7, 3, 3, 2) | 1.00 [1.00 to 6.02] | 2.00 [2.00 to 3.00] | 1.03 [1.00 to 2.33] | 1.97 [0.917 to 4.00] | 1.07 [1.00 to 2.00] | 1.00 [0.333 to 4.00] | 2.00 [1.00 to 4.00] | 2.50 [1.00 to 4.00]
  Cycle 1 Day 1 (N=5, 3, 3, 6, 6, 3, 4, 2) | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 4.00] | 1.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 1.00 [1.00 to 2.02] | 2.00 [2.00 to 4.05] | 1.50 [1.00 to 6.00] | 1.00 [1.00 to 1.00]

18. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for PD-0325901 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm A
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
hr
  Cycle 0 Day -7 (N=5, 1, 1) | 1.00 [1.00 to 4.00] | 2.00 [2.00 to 2.00] | 1.92 [1.92 to 1.92]
  Cycle 1 Day 12 (N=4, 1, 1) | 1.00 [1.00 to 1.02] | 1.00 [1.00 to 1.00] | 4.00 [4.00 to 4.00]

19. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for PF-04691502 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm A
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
hr
  Cycle 0 Day -7 (N=5, 1, 1) | 1.00 [1.00 to 6.00] | 1.00 [1.00 to 1.00] | 1.90 [1.90 to 1.90]
  Cycle 1 Day 12 (N=4, 1, 1) | 2.00 [1.02 to 2.00] | 0.00 [0.00 to 0.00] | 2.00 [2.00 to 2.00]

20. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) for PF-04691502 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm B
Time Frame: as for outcome 14
Population: as for outcome 10
Measure: Median (Full Range); unit: hr
Arm/Group | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1)
Number analyzed (Participants) | 7 | 7
hr
  Cycle 0 Day -7 (N=7, 7) | 2 [1 to 8] | 1.07 [1 to 4.13]
  Cycle 1 Day 12 (N=7, 5) | 2 [1 to 4] | 2.03 [1.02 to 6]

21. Secondary Outcome: Terminal Elimination Half Life (t½) for PF-05212384 on Cycle 1 Day 2 and Day 16 for Arm C
Time Frame: Cycle 1 Day 2 and Cycle 1 Day 16: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2)
Number analyzed (Participants) | 1 | 5 | 3 | 25
hr
  Cycle 1 Day 2 (N=1, 5, 3, 25) | 24.5 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 32.14 (1.3334) | 29.23 (7.1066) | 32.16 (4.5154)
  Cycle 1 Day 16 (N=1, 5, 3, 20) | 33.3 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 37.98 (5.5603) | 34.50 (8.4256) | 35.10 (3.3067)

22. Secondary Outcome: Terminal Elimination Half Life (t½) for PF-05212384 on Cycle 0 Day -14 and Cycle 1 Day 15 for Arm D
Time Frame: Day -14 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 3 | 3 | 6 | 6 | 3 | 4 | 2
hr
  Cycle 0 Day -14 (N=5, 3, 3, 6, 6, 3, 4, 2) | 24.62 (3.2306) | 27.37 (6.4748) | 30.77 (6.4933) | 25.85 (4.1530) | 29.35 (5.5121) | 29.63 (3.7072) | 27.05 (4.6651) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 24.6 and 24.8 hr, respectively.
  Cycle 1 Day 15 (N=3, 3, 4, 6, 3, 1, 3, 1) | 35.90 (4.8816) | 39.30 (10.678) | 41.25 (6.2303) | 34.43 (8.5383) | 40.20 (5.8643) | 37.0 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. | 33.30 (0.96437) | 37.0 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP.

23. Secondary Outcome: Terminal Elimination Half Life (t½) for PD-0325901 on Cycle 0 Day -7 for Arm A
Time Frame: Cycle 0 Day -7: Pre-dose and 1, 2, 4, 6, 8, 24, and 72 hours post-dose.
Population: Enrolled participants treated who had at least 1 of the pharmacokinetic (PK) parameters of interest estimated.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
hr | 13.92 (4.2260) | 18.3 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 25.7 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

24. Secondary Outcome: Terminal Elimination Half Life (t1/2) for PF-04691502 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm A
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
hr
  Cycle 0 Day -7 (N=5, 1, 1) | 9.374 (1.3243) | 12.4 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 11.5 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.
  Cycle 1 Day 12 (N=4, 0, 0) | 8.968 (1.5366) | NA (NA) — N = 0. | NA (NA) — N = 0.

25. Secondary Outcome: Terminal Elimination Half Life (t1/2) for PF-04691502 on Cycle 0 Day -7 and Cycle 1 Day 12 for Arm B
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1)
Number analyzed (Participants) | 6 | 7
hr
  Cycle 0 Day -7 (N=6, 7) | 13.13 (2.2879) | 13.06 (2.6589)
  Cycle 1 Day 12 (N=3, 1) | 8.597 (1.2726) | 8.97 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

26. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-05212384 on Cycle 1 Day 2 and Cycle 1 Day 16 for Arm C
Time Frame: Cycle 1 Day 2 and Cycle 1 Day 16: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2)
Number analyzed (Participants) | 3 | 6 | 4 | 31
ng*hr/mL
  Cycle 1 Day 2 (N=2, 6, 4, 30) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 7410 and 10500 ng*hr/mL, respectively. | 7487 (41) | 10530 (44) | 9485 (43)
  Cycle 1 Day 16 (N=3, 6, 4, 28) | 8819 (71) | 8243 (25) | 11170 (53) | 10890 (38)

27. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-05212384 on Cycle 0 Day -14 and Cycle 1 Day 15 for Arm D
Time Frame: Cycle 0 Day -14 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
ng*hr/mL
  Cycle 0 Day -14 (N=7, 3, 4, 7, 6, 3, 4, 2) | 7627 (46) | 10250 (21) | 14850 (31) | 12590 (27) | 14280 (24) | 13840 (47) | 9619 (22) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 14900 and 18800 ng*hr/mL, respectively.
  Cycle 1 Day 15 (N=5, 3, 4, 6, 5, 1, 4, 1) | 12070 (36) | 12130 (1) | 19970 (25) | 13390 (21) | 21170 (36) | 15200 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. | 12610 (25) | 20800 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP.

28. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PD-0325901 on Cycle 0 Day -7 for Arm A
Time Frame: Cycle 0 Day -7: Pre-dose and 1, 2, 4, 6, 8, 24, and 72 hours post-dose.
Population: Enrolled participants treated who had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
ng*hr/mL | 1479 (23) | 2030 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 941 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

29. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-04691502 on Cycle 0 Day -7 for Arm A
Time Frame: as for outcome 13
Population: Enrolled participants treated who had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
ng*hr/mL | 474.5 (29) | 933 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 688 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

30. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-04691502 on Cycle 0 Day -7 for Arm B
Time Frame: as for outcome 13
Population: Enrolled participants treated who had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1)
Number analyzed (Participants) | 7 | 7
ng*hr/mL | 588.4 (49) | 1001 (35)

31. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-05212384 on Cycle 1 Day 2 and Cycle 1 Day 16 for Arm C
Time Frame: Cycle 1 Day 2 and Cycle 1 Day 16: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2)
Number analyzed (Participants) | 3 | 6 | 4 | 31
ng*hr/mL
  Cycle 1 Day 2 (N=1, 5, 3, 25) | 7540 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 7968 (41) | 9277 (48) | 10070 (42)
  Cycle 1 Day 16 (N=1, 5, 3, 20) | 5870 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 8627 (26) | 9174 (17) | 10610 (37)

32. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-05212384 on Cycle 0 Day -14 and Cycle 1 Day 15 for Arm D
Time Frame: Cycle 0 Day -14 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 4, 6, 8, 24, 72, and 120 hours post-dose.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
ng*hr/mL
  Cycle 0 Day -14 (N=5, 3, 3, 6, 6, 3, 4, 2) | 6353 (40) | 10460 (20) | 14880 (39) | 12600 (29) | 14620 (23) | 14230 (46) | 9766 (22) | NA (NA) — For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. Individual values of these 2 participants were 15100 and 19100 ng*hr/mL, respectively.
  Cycle 1 Day 15 (N=3, 3, 4, 6, 3, 1, 3, 1) | 10430 (33) | 12460 (2) | 20440 (26) | 13770 (20) | 23730 (39) | 15500 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP. | 13320 (27) | 21300 (NA) — Individual value is reported. For arms with <3 participants with reportable values, data summary statistics were not calculated per standard practice and as specified in the SAP.

33. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PD-0325901 on Cycle 0 Day -7 for Arm A
Time Frame: Cycle 0 Day -7: Pre-dose and 1, 2, 4, 6, 8, 24, and 72 hours post-dose.
Population: Enrolled participants treated who had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
ng*hr/mL | 1599 (26) | 2140 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 1060 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

34. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-04691502 on Cycle 0 Day -7 for Arm A
Time Frame: as for outcome 13
Population: Enrolled participants treated who had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 1
ng*hr/mL | 523.9 (21) | 950 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values. | 697 (NA) — Individual value is reported. Summary statistics are not presented if fewer than 3 subjects have reportable parameter values.

35. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-04691502 on Cycle 0 Day -7 for Arm B
Time Frame: as for outcome 13
Population: Enrolled participants treated who had at least 1 of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1)
Number analyzed (Participants) | 6 | 7
ng*hr/mL | 705.0 (41) | 1028 (36)

36. Secondary Outcome: Number of Participants With Increase From Baseline in QT Interval
Description: Electrocardiogram (ECG) measurements (an average of the triplicate measurements) were used for the statistical analysis and all data presentations. QT intervals were corrected for heart rate (QTc) using Bazett's Formula (QTcB) and Fridericia's Formula (QTcF) .
Time Frame: Baseline, Cycle 1 Day 2 for Arms C and D, Cycle 1 Day 15 for Arm D, and Cycle 1 Day 16 for Arm C, Day 2 in Arm C and Day 1 in Arm D for subsequent cycles, up to End of Treatment (within 28 days of last treatment administration)
Population: All participants enrolled in the study having at least one ECG assessment after receiving study drug for the respective arm.
Measure: Number; unit: participants
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 30 | 7 | 3 | 3 | 7 | 5 | 3 | 4 | 2
participants
  Maximum QTcB Interval Increase <30msec | 4 | 0 | 1 | 7 | 7 | 2 | 5 | 4 | 28 | 7 | 2 | 2 | 6 | 4 | 3 | 3 | 2
  MaximumQTcB Interval Increase >=30to<60msec | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
  Maximum QTcB Interval Increase >=60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTcF Interval Increase <30 msec | 5 | 0 | 1 | 7 | 5 | 2 | 5 | 3 | 24 | 6 | 3 | 2 | 6 | 5 | 3 | 4 | 2
  MaximumQTcF Interval Increase >=30 to<60msec | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 6 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Maximum QTcF Interval Increase >=60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: Number of Participants With Maximum Post-dose QT Interval Corrected
Description: Electrocardiogram (ECG) measurements (an average of the triplicate measurements) were used for the statistical analysis and all data presentations. QT intervals were corrected for heart rate (QTc) using Bazett's Formula (QTcB) and Fridericia's Formula (QTcF).
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Number; unit: participants
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 7 | 3 | 6 | 4 | 31 | 7 | 3 | 4 | 7 | 7 | 3 | 4 | 2
participants
  Maximum QTcB Interval <450 msec | 2 | 0 | 1 | 4 | 3 | 2 | 4 | 1 | 22 | 2 | 3 | 3 | 2 | 4 | 3 | 2 | 1
  Maximum QTcB Interval 450 to <=480 msec | 3 | 0 | 0 | 3 | 4 | 1 | 2 | 3 | 5 | 5 | 0 | 1 | 5 | 1 | 0 | 1 | 0
  Maximum QTcB Interval >480 to <=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
  Maximum QTcB Interval >500 msec | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Maximum QTcF Interval <450 msec | 4 | 0 | 1 | 7 | 3 | 3 | 6 | 2 | 24 | 6 | 3 | 4 | 6 | 5 | 3 | 2 | 1
  Maximum QTcF Interval 450 to <=480 msec | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 5 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  Maximum QTcF Interval >480 to <=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Maximum QTcF Interval >500 msec | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR)
Description: CR was defined as the disappearance of all target lesions with the exception of nodal disease and all target nodes must decrease to normal size (short axis <10 mm). PR was defined as at least a 30% decrease in the sum of the longest diameters of the targeted lesions.
Time Frame: Baseline, every 8 weeks in Cycle 3 and subsequent cycles, until progression of disease was documented.
Population: All participants who started treatment on the assigned arm and had an adequate baseline tumor assessment.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 7 | 6 | 3 | 6 | 4 | 30 | 7 | 3 | 3 | 7 | 7 | 3 | 4 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0 | 33.3 [0.8 to 90.6] | 0 [0.0 to 45.9] | 0 [0.0 to 60.2] | 3.3 [0.1 to 17.2] | 0 [0.0 to 41.0] | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8] | 28.6 [3.7 to 71.0] | 14.3 [0.4 to 57.9] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 84.2]

39. Secondary Outcome: Progression-Free Survival (PFS) (Stage 2)
Description: Progression-free survival (PFS) was the time from first dose to date of first documentation of progression or death due to any cause.
Time Frame: Baseline, every 8 weeks in Cycle 3 and subsequent cycles, until progression of disease was documented.
Population: All participants who started treatment on the assigned arm and had an adequate baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-05212384+Irinotecan: Arm C2 (Stage 2)
Number analyzed (Participants) | 30
months | 2.8 [1.7 to 3.7]

40. Secondary Outcome: Ratio to Baseline in Serum Glucose Level at End of Treatment for Arm B, Arm C, and Arm D
Time Frame: Baseline, Cycle 1 Days 2, 15, 22, and 23, Cycle 2 Days 1 and 16, Day 1 in Cycle 3 and subsequent cycles, and EOT (within 28 days after last treatment administration)
Population: All enrolled participants who started treatment and had baseline and on treatment serum biomarker samples (glucose, insulin, or other serum biomarkers) successfully analyzed for at least one of the biomarkers.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 5 | 2 | 5 | 3 | 25 | 5 | 3 | 2 | 6 | 5 | 3 | 4 | 1
ratio | 0.974 (0.0864) | 1.015 (0.1935) | NA (NA) — Arm C1 for Stage 1 had 2 participants with data at End of treatment and were not summarized. The individual values were 1.305 and 1.293. | 1.011 (0.1165) | NA (NA) — Arm C3 for Stage 1 had 3 participants with data at End of treatment and were not summarized. The individual values were 0.64, 1.262, and 1.093. | 1.111 (0.2895) | 1.212 (0.3284) | NA (NA) — Arm D0A for Stage 1 had 3 participants with data at End of treatment and were not summarized. The individual values were 0.708 , 0.973 and 1.024. | NA (NA) — Arm D0B for Stage 1 had 2 participants with data at End of treatment and were not summarized. The individual values were 0.956 and 1.104. | 0.966 (0.1904) | 1.13 (0.3886) | NA (NA) — Arm D1B for Stage 1 had 3 participants with data at End of treatment and were not summarized. The individual values were 1.641,1.198 and 0.947. | NA (NA) — Arm D2 for Stage 1 had 4 participants with data at End of treatment and were not summarized. The individual values were 0.93, 0.74, 1.113 and 0.817. | NA (NA) — Arm D2A for Stage 1 had 1 participants with data at End of treatment and were not summarized. The individual values was 0.783.

41. Secondary Outcome: Ratio to Baseline in Serum Insulin Level at End of Treatment for Arm B, Arm C, and Arm D
Time Frame: as for outcome 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 4 | 6 | 2 | 5 | 3 | 22 | 4 | 3 | 1 | 5 | 4 | 3 | 4 | 1
ratio | NA (NA) — Arm B1 for Stage 1 had 4 participants with data at End of treatment and were not summarized. The individual values were 0.412, 2.2, 1, 0.973. | 1.628 (1.888) | NA (NA) — Arm C1 for Stage 1 had 2 participants with data at End of treatment and were not summarized. The individual values were 1.528 and 1.14. | 2.178 (2.3194) | NA (NA) — Arm C3 for Stage 1 had 3 participants with data at End of treatment and were not summarized. The individual values were 0.244, 0.769, 0.552. | 1.699 (2.0031) | NA (NA) — Arm D0 for Stage 1 had 4 participants with data at End of treatment and were not summarized. The individual values were 0.833, 5.143, 0.979, 0.744. | NA (NA) — Arm D0A for Stage 1 had 3 participants with data at End of treatment and were not summarized. The individual values were 0.374, 0.905, 0.736. | NA (NA) — Arm D0B for Stage 1 had 1 participant with data at End of treatment and was not summarized. The individual value was 1.434. | 2.233 (2.3617) | NA (NA) — Arm D1A for Stage 1 had 4 participants with data at End of treatment and were not summarized. The individual values were2.026, 0.665, 0.32, 4.404. | NA (NA) — Arm D1B for Stage 1 had 3 participants with data at End of treatment and were not summarized. The individual values were 2.116, 1.187, 1.172. | NA (NA) — Arm D2 for Stage 1 had 4 participants with data at End of treatment and were not summarized. The individual values were 0.403, 0.281, 3.293, 3.776. | NA (NA) — Arm D2A for Stage 1 had 1 participant with data at End of treatment and was not summarized. The individual value was 0.083.

42. Secondary Outcome: Ratio to Baseline in Serum Glucose Level at Cycle 2 Day 16 for Arm A
Time Frame: as for outcome 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 0
ratio | 0.965 (0.2697) | NA (NA) — Arm A2 for Stage 1 had only 1 participant with data at Cycle 2 Day 16 and was not summarized. The individual value for the 1 participant was 1.035. |

43. Secondary Outcome: Ratio to Baseline in Serum Insulin Level at Cycle 2 Day 16 for Arm A
Time Frame: as for outcome 40
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1)
Number analyzed (Participants) | 5 | 1 | 0
ratio | 0.652 (0.3622) | NA (NA) — Arm A2 for Stage 1 had only 1 participant with data at Cycle 2 Day 16 and was not summarized. The individual value for the 1 participant was 0.972. |

44. Secondary Outcome: Number of Participants With Expression of Genes Relating to Phosphatidylinositol 3 Kinase (PI3K), Mitogen Activated Protein Kinase (MAPK) and/or Wingless-Type Mouse Mammary Tumor Virus Integration Site Family Member (Wnt) Pathway Signaling
Description: Number of participants with expression of genes relating to PI3K, MAPK and/or Wnt pathway signaling (kirsten rat sarcoma 2 viral oncogene homolog [KRAS] and PTEN protein). Biopsies were obtained at baseline and Cycle 1 Day 23. Biomarker evaluation was performed on these biopsies.
Time Frame: Baseline and Cycle 1 Day 23.
Population: All enrolled participants who started treatment and had baseline tumor tissues successfully analyzed for at least one of the biomarkers.
Measure: Number; unit: participants
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+ PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+PD-0325901: Arm D1B (Stage 1) | PF-05212384+PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Number analyzed (Participants) | 5 | 1 | 1 | 6 | 7 | 3 | 5 | 4 | 24 | 4 | 2 | 3 | 6 | 7 | 3 | 2 | 1
participants
  KRAS mutation | 4 | 1 | 1 | 0 | 3 | 0 | 2 | 1 | 10 | 2 | 1 | 2 | 4 | 6 | 2 | 1 | 1
  PTEN tumor manual score | 4 | 1 | 1 | 5 | 6 | 3 | 5 | 4 | 24 | 4 | 2 | 3 | 6 | 7 | 2 | 2 | 1
  PTEN stroma manual score | 4 | 1 | 1 | 5 | 6 | 3 | 4 | 4 | 24 | 4 | 2 | 3 | 6 | 7 | 2 | 2 | 1

45. Secondary Outcome: Duration of Response (Stage 2)
Description: Duration of response was to be calculated for participants with an objective response. Duration of PR or CR was the time from start date (date of first documentation of PR or CR) to date of first documentation of objective progression or death. CR: disappearance of a target lesions. PR: at least 30% decrease in the sum of diameters of target lesions.
Time Frame: Baseline, every 8 weeks in Cycle 3 and subsequent cycles, until until progression of disease was documented.
Population: There was only 1 participant in Arm C1 and 1 in Arm C2 with a response, therefore summary statistics were not calculated for this endpoint.
Arm/Group | PF-05212384+Irinotecan: Arm C2 (Stage 2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to End of Treatment (EOT) (within 28 days after last treatment administration).
Groups:
- PF-05212384+PD-0325901: Arm D0A (Stage 1): Single intravenous dose of PF-05212384 130 mg in lead-in period (Day 14 prior to Cycle 1 day 1) followed by intravenous doses of PF-05212384 130 mg on Days 1, 8, 15 and 22. Single oral dose of PF 0325901 2 mg capsule in lead-in period (Day 7 to Day 1 prior to Cycle 1 Day 1), followed by PF 0325901 2 mg capsule orally twice daily continuously on Days 2-12 and 16-26 of each cycle until participants experienced unacceptable toxicity, disease progression, withdrawal from the study, or death.
Arm/Group | PF-04691502+PF-0325901: Arm A1 (Stage1) | PF-04691502+PF 0325901: Arm A2 (Stage1) | PF-04691502+PF 0325901: Arm A4 (Stage1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) | PF-04691502+Irinotecan: Arm B2 (Stage 1) | PF-05212384+Irinotecan: Arm C1 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 1) | PF-05212384+Irinotecan: Arm C3 (Stage 1) | PF-05212384+Irinotecan: Arm C2 (Stage 2) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) | PF-05212384+PD-0325901: Arm D0A (Stage 1) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) | PF-05212384+ PD-0325901: Arm D1B (Stage 1)) | PF-05212384+ PD-0325901: Arm D2 (Stage 1) | PF-05212384+ PD-0325901: Arm D2A (Stage 1)
Serious Adverse Events (participants affected / at risk) | 2/5 | 1/1 | 1/1 | 2/7 | 5/7 | 0/3 | 0/6 | 2/4 | 5/31 | 3/7 | 1/3 | 2/4 | 4/7 | 1/7 | 0/3 | 1/4 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1 | 1/1 | 7/7 | 7/7 | 3/3 | 6/6 | 4/4 | 31/31 | 7/7 | 3/3 | 4/4 | 7/7 | 7/7 | 3/3 | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04691502+PF-0325901: Arm A1 (Stage1) (N=5) | PF-04691502+PF 0325901: Arm A2 (Stage1) (N=1) | PF-04691502+PF 0325901: Arm A4 (Stage1) (N=1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) (N=7) | PF-04691502+Irinotecan: Arm B2 (Stage 1) (N=7) | PF-05212384+Irinotecan: Arm C1 (Stage 1) (N=3) | PF-05212384+Irinotecan: Arm C2 (Stage 1) (N=6) | PF-05212384+Irinotecan: Arm C3 (Stage 1) (N=4) | PF-05212384+Irinotecan: Arm C2 (Stage 2) (N=31) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) (N=7) | PF-05212384+PD-0325901: Arm D0A (Stage 1) (N=3) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) (N=4) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) (N=7) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) (N=7) | PF-05212384+ PD-0325901: Arm D1B (Stage 1)) (N=3) | PF-05212384+ PD-0325901: Arm D2 (Stage 1) (N=4) | PF-05212384+ PD-0325901: Arm D2A (Stage 1) (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-04691502+PF-0325901: Arm A1 (Stage1) (N=5) | PF-04691502+PF 0325901: Arm A2 (Stage1) (N=1) | PF-04691502+PF 0325901: Arm A4 (Stage1) (N=1) | PF-04691502+Irinotecan: Arm B1 (Stage 1) (N=7) | PF-04691502+Irinotecan: Arm B2 (Stage 1) (N=7) | PF-05212384+Irinotecan: Arm C1 (Stage 1) (N=3) | PF-05212384+Irinotecan: Arm C2 (Stage 1) (N=6) | PF-05212384+Irinotecan: Arm C3 (Stage 1) (N=4) | PF-05212384+Irinotecan: Arm C2 (Stage 2) (N=31) | PF-05212384+ PD-0325901: Arm D0 (Stage 1) (N=7) | PF-05212384+PD-0325901: Arm D0A (Stage 1) (N=3) | PF-05212384+ PD-0325901: Arm D0B (Stage 1) (N=4) | PF-05212384+ PD-0325901: Arm D1 (Stage 1) (N=7) | PF-05212384+ PD-0325901: Arm D1A (Stage 1) (N=7) | PF-05212384+ PD-0325901: Arm D1B (Stage 1)) (N=3) | PF-05212384+ PD-0325901: Arm D2 (Stage 1) (N=4) | PF-05212384+ PD-0325901: Arm D2A (Stage 1) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 7 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 0 | 3 | 3 | 1 | 2 | 3 | 17 | 1 | 1 | 2 | 3 | 5 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 5 | 5 | 3 | 3 | 2 | 19 | 1 | 2 | 1 | 3 | 5 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 6 | 2 | 1 | 1 | 0 | 4 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 6 | 4 | 1 | 3 | 2 | 14 | 2 | 1 | 2 | 3 | 5 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 1 | 10 | 2 | 2 | 2 | 0 | 1 | 1 | 2 | 0
Fatigue (General disorders) | 3 | 1 | 0 | 3 | 3 | 2 | 2 | 2 | 9 | 3 | 1 | 0 | 4 | 5 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 6 | 1 | 0 | 1 | 2 | 3 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 | 4 | 2 | 1 | 3 | 12 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 7 | 2 | 0 | 1 | 3 | 1 | 1 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 12 | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 7 | 2 | 1 | 3 | 3 | 3 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 3 | 2 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 5 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 6 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 5 | 1 | 1 | 1 | 4 | 3 | 1 | 1 | 2
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1/13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 3 | 4 | 2 | 0 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 1 | 2 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fistula discharge (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Choluria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ejaculation failure (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated prematurely for strategic reasons based on an internal portfolio prioritization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.